CLINICAL TRIAL: NCT07170410
Title: Sigmoid Colon Volvulus in the Population Groups of Sohag
Brief Title: Sigmoid Colon Volvulus in Sohag
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Hesham Mohamed Hashem, General surgury resident at sohag university hospital, Sohag University
Other Study IDs: Soh-Med--25-8-9MS
Record Dates: First submitted 2025-09-05; First posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Sigmoid Volvulus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary goal of this study observational is to highlight the paradigm of sigmoid colon volvulus as a cause of large intestinal obstruction in young age groups in addition to the elderly for early diagnosis and thus avoiding complications.

ELIGIBILITY:
Inclusion Criteria: All patients with a clinical diagnosis of Sigmoid colon volvulus males or females, of any age, -

Exclusion Criteria:.Sigmoid mass, Sigmoidopexy, pelvic inflammatory disease, TB pelvis, abdomen, Any stoma (colostomy, Iliostomy).

-

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: population groups of Sohag
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
highlight the paradigm of SV as a cause of large intestinal obstruction in young age groups in addition to the elderly | 3 years
  highlight the paradigm of SV as a cause of large intestinal obstruction in young age groups in addition to the elderly

IPD SHARING:
Plan to Share IPD: Undecided